CLINICAL TRIAL: NCT07250386
Title: A Clinical Study to Evaluate the Safety and Efficacy of CEA-Targeted Chimeric Antigen Receptor T (CAR-T) Cells in Patients With CEA-Positive Advanced Malignant Solid Tumors
Brief Title: A Study of CEA-Targeted CAR-T Therapy in Patients With CEA-Positive Advanced Solid Tumors
Acronym: PBC102
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0883
Record Dates: First submitted 2025-09-24; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer); Breast Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Two experimental cohorts by infusion route - intravenous (IV) and intrathoracic (IT). Each cohort conducts sequential dose escalation using an enhanced 3+3 design (3 dose levels; 3-6 participants per level depending on DLTs), followed by optional dose expansion at 1-2 selected dose levels. The two route cohorts may run in parallel operationally, but enrollment within each cohort proceeds sequentially per the dose-escalation scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 2-6x10^5 cells/kg
  Interventions: Biological: CEA-targeted CAR-T (Intravenous)
- Intrapleural infusion of CEA-targeted CAR-T (Experimental): Infusion of CEA-targeted CAR-T cells by dose of 2-6x10^5 cells/kg
  Interventions: Biological: CEA-targeted CAR-T (Intrapleural)

INTERVENTIONS:
Biological: CEA-targeted CAR-T (Intravenous) — Administration method: intravenous infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion
  Arms: Intravenous of CEA-targeted CAR-T
Biological: CEA-targeted CAR-T (Intrapleural) — Administration method: intrapleural infusion. Subjects will receive conditioning therapy by Fludarabine and Cyclophosphamide before cell infusion
  Arms: Intrapleural infusion of CEA-targeted CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalating + dose-expansion clinical study, aiming to evaluate the safety and efficacy of CEA-targeted CAR-T cell preparations, and to preliminarily observe the study drug in CEA-positive advanced malignant tumors. The pharmacokinetic characteristics of CAR-T cell preparations for the treatment of patients with CEA-positive advanced malignancies were obtained and the recommended dose and infusion schedule.

DETAILED DESCRIPTION:
According to the different infusion methods, patients will be assigned to two parallel subgroups: intravenous infusion, intrapleural infusion.

Within each subgroup, the study is conducted in two sequential parts:

1. .Part A (dose-escalation): escalation begins at the lowest dose level; 3-6 subjects are enrolled at each dose level;
2. .Part B (dose-expansion): additional subjects are treated at the recommended dose identified in Part A to further evaluate safety and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older, of any gender.
2. Histologically or cytologically confirmed advanced, metastatic, or recurrent solid tumors, including non-small cell lung cancer and breast cancer.
3. Disease progression or intolerance after at least second-line standard therapy, including but not limited to surgery, chemotherapy, radiotherapy, targeted therapy, or immunotherapy.
4. CEA positivity confirmed by immunohistochemistry (IHC) in tumor samples within 3 months of screening (clear membrane staining, with positivity rate ≥10%). If the IHC result is more than 3 months old, serum CEA must be above 10 ng/mL.
5. At least one evaluable lesion according to RECIST 1.1, with a longest diameter of ≥10 mm for non-lymph node lesions and a shortest diameter of ≥15 mm for lymph node lesions. Malignant pleural effusion is acceptable for the chest infusion subgroup.
6. For patients with malignant pleural effusion, accurate volume assessment of pleural effusion by imaging (CT or MRI) and cytological or thoracoscopic biopsy confirmation of malignant pleural effusion.
7. ECOG performance status of 0-2.
8. Life expectancy of 12 weeks or more.
9. No serious psychiatric disorders.
10. The following organ function criteria should be met unless otherwise specified:

    1. Hematology: White blood cell count >2.0×10^9/L, neutrophils >1.0×10^9/L, lymphocytes >0.5×10^9/L, platelets >50×10^9/L, hemoglobin >80 g/L.
    2. Cardiac function: Echocardiography showing ejection fraction ≥50%, with no significant abnormalities on ECG.
    3. Renal function: Serum creatinine ≤2.0×ULN.
    4. Liver function: ALT and AST ≤3.0×ULN (≤5.0×ULN for those with liver tumor infiltration).
    5. Total bilirubin ≤2.0×ULN.
    6. Oxygen saturation >92% without supplemental oxygen.
11. Eligible for single or venous blood collection with no contraindications to cell collection.
12. Consent to use a reliable and effective method of contraception for 1 year after CAR-T cell infusion (excluding the rhythm method).
13. The participant or their authorized guardian agrees to participate in the clinical trial and signs the informed consent form (ICF), indicating an understanding of the trial's purpose and procedures.

Exclusion Criteria:

1. Clinical symptoms of CNS metastasis or meningeal metastasis at screening, or other evidence suggesting that CNS metastasis or meningeal metastasis is uncontrolled, as determined by the investigator.
2. Participation in other clinical trials within 4 weeks prior to screening.
3. Receipt of a live attenuated vaccine within 4 weeks prior to screening.
4. Receipt of chemotherapy, targeted therapy, or other experimental drugs within 14 days or at least 5 half-lives (whichever is shorter) prior to screening.
5. Active or uncontrolled infection requiring systemic treatment.
6. Tumor compression of the trachea or major blood vessels, with significant risk as assessed by the investigator.
7. History of any of the following cardiac diseases:

   1. New York Heart Association (NYHA) Class III or IV congestive heart failure.
   2. Myocardial infarction or coronary artery bypass grafting (CABG) within 6 months prior to screening.
   3. Clinically significant ventricular arrhythmias or unexplained syncope (except those caused by vasovagal or dehydration).
   4. History of severe non-ischemic cardiomyopathy.
8. Active autoimmune disease or other conditions requiring long-term immunosuppressive therapy.
9. History of or concurrent untreated malignancies within 3 years, except for basal cell carcinoma or in situ cervical cancer.
10. Positive for HBsAg or HBcAb with HBV DNA levels above the normal range, HCV antibody positive with HCV RNA levels above the normal range, HIV antibody positive, or positive for syphilis.
11. Pregnant or breastfeeding women.
12. Any other condition that the investigator deems unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of CAR-T cell preparations in the treatment of CEA-positive advanced malignancies [Safety and Tolerability] | From infusion through Month 3
  Incidence of adverse events during the study, evaluated per the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and American Society for Transplantation and Cellular Therapy (ASTCT) criteria
Obtained the recommended dose and infusion regimen of CAR-T cells for the treatment of patients with CEA-positive advanced malignancies [Safety and Tolerability] | From infusion through Month 3
  Dose-limiting toxicity after CEA CAR-T cell infusion

SECONDARY OUTCOMES:
Assessing disease control(DCR) rates of CAR-T cell preparations in CEA-positive advanced malignancies [Effectiveness] | From infusion through Month 3
  DCR: The proportion of subjects who achieved CR, PR, SD after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Objective response rate (ORR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  Objective response rate includes：The proportion of subjects who achieved CR, PR after CAR-T infusion accounted for all treated subjects (Assessed based on RECIST criteria)，the minimum value is 0%，maximum value is 100%, and higher scores mean a better outcome.
Duration of Response (DOR) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death(Assessed based on RECIST criteria)
Progress-free survival(PFS) of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  PFS will be assessed from the first CEA-CAR-T cell infusion to death from any cause or the first assessment of progression(Assessed based on RECIST criteria)
Overall survival(OS)of CEA CAR-T treatment in patients with CEA-positive advanced malignancies [Effectiveness] | 2 years
  OS will be assessed from the first CEA-CAR-T cell infusion to death from any cause (Assessed by investigators based on IRECIST criteria)
To evaluate the efficacy of CAR-T cell preparations in CEA-positive advanced malignancies【Effectiveness】 | 2 years
  Changes in serum tumor marker levels: CEA, CA-125, etc.
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  Cmax: maximum observed level of circulating CAR-T cells in peripheral blood after infusion
To characterize the in-vivo cellular kinetics of CAR-T cells【pharmacokinetics】 | From infusion through Month 3
  To determine the time to maximum observed level of circulating CAR-T cells (Tmax)
To characterize the in-vivo cellular kinetics of CAR [T cells#pharmacokinetics] | From infusion through Month 3
  To estimate AUC0-28d and AUC0-90d for circulating CAR-T cells

OTHER OUTCOMES:
Change in Residual Tumor Cells after CEA CAR-T Therapy | 2 years
  Assess changes in residual tumor cells before and after CEA CAR-T therapy to identify potential biomarkers associated with therapeutic response
Change in CEA Expression after CEA CAR-T Therapy | 2 years
  Assess changes in CEA expression before and after CEA CAR-T therapy to identify potential biomarkers associated with therapeutic response
Change in Tumor-Infiltrating Immune Cells after CEA CAR-T Therapy | 2 years
  Assess changes in tumor-infiltrating immune cells (e.g., T cells, NK cells, macrophages) before and after CEA CAR-T therapy to identify potential biomarkers associated with therapeutic response
Change in Multi-omics Profiles after CEA CAR-T Therapy | 2 years
  Assess changes in multi-omics profiles (e.g., genomics, transcriptomics, proteomics) before and after CEA CAR-T therapy to identify potential biomarkers associated with therapeutic response

CONTACTS AND LOCATIONS:
Overall Officials: Fuming Qiu, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Junqiang Fan, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No